CLINICAL TRIAL: NCT03963115
Title: Can Epinephrine Coated Syringe for Subcutaneous Immunotherapy (SCIT) Reduce Large Local Reaction?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Professor, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 393/2561(EC3)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Injection Reactions Site; Systemic Reactions
Keywords: Large local reaction; adrenaline, epinephrine
MeSH Terms: conditions — Injection Site Reaction | interventions — Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, crossover trial with epinephrine coated syringe before injected and placebo was done in each visit in patients who developed large local reactions after subcutaneous immunotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were randomly assigned to receive either epinephrine or normal saline (placebo) coated syringe for SCIT by a block of 4 randomization. These syringes were used to draw allergen extracts. The syringes for the second visit were coated with different agents from the first visit in the same patients. One investigator (K.B.) generated the allocation sequence and prepared the coated syringes. The physicians who drew and injected the allergen shots and the patients were blinded to the assignment from the beginning to the end of the interventions. Interventions were decoded at the end of the study by K.B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coated syringe with epinephrine (Active Comparator): Epinephrine was coated syinge before drawing the allergen to filled in.
  Interventions: Drug: Epinephrine or normal saline
- placebo (Placebo Comparator): Normal saline was coated syinge before drawing the allergen to filled in.
  Interventions: Drug: Epinephrine or normal saline

INTERVENTIONS:
Drug: Epinephrine or normal saline — epinephreine or normal saline coated syringe before drawing allergen for injection.
  Other Names: Adrenaline or normal saline

SUMMARY:
Allergen immunotherapy is effective in the management of allergic asthma, allergic rhinitis/conjunctivitis, and stinging insect hypersensitivity. The most common side effect of subcutaneous allergen specific immunotherapy (SCIT) is local reactions (LR). Although some studies indicated that LR did not predict systemic reaction (SR), patients with higher frequency of large local reaction (LLR) were reported to have higher risk for SR. Epinephrine may decrease LLR due to its vasoconstrictive effect . The objective of this study was to compare the size of LLR in patients receiving SCIT with epinephrine or normal saline coated syringe. The patients who complained of frequent LLR despite pre-medication and local treatment were recruited.

DETAILED DESCRIPTION:
Allergen immunotherapy (AIT) is an immune mediated treatment which modifies T helper (Th) 2-directed response through the interplay between regulatory T and B cells, blocking IgG4 antibodies and tissue effector-mediated mechanisms. Aeroallergen immunotherapy is recommended for patients with allergic rhinitis, allergic conjunctivitis or allergic asthma whose symptoms were not adequately controlled by antigen avoidance and pharmacotherapy. AIT could reduce symptoms and medication usage in respiratory allergy. In children, AIT prevented the progression from allergic rhinitis to asthma and prevented new onset of allergen sensitization in monosensitized patients. The administration of allergen by subcutaneous injection (SCIT) is a common practice among allergists.

The benefits of SCIT must be weighed against the risks of side effects which can be mild or life threatening. Adverse allergic reactions to SCIT were classified as either local (LR) or systemic reactions (SR).6 Large local reactions (LLR) are defined as erythema and/or swelling (> 25 mm) at the site of injection. The timing of adverse reactions were categorized into immediate (occurring within 30 min) and late reactions (occurring > 30 min after injection). LR associated with SCIT ranged from 26-72% of patients and 0.7-4% of injections. SR were reported to occurred in 3.7% of patients and 0.3% of injection. Recent prospective study in pediatric patients who received SCIT showed immediate LR in 54.6%, delayed LR in 56.1%, immediate SR in 2.2% and delayed SR in 7.4% of the patients. Severe SR were seen in 0.03% of all treatments which appeared within 30 minutes after the injections. The author concluded that children had similar rates of LR compared to adult patients but had lower rates of severe SR.

Several studies indicated that individual LR did not predict subsequent SR. The rate of SR were not change despite the dose adjustment after a LR. However, patients with greater frequency of LLR might be at an increased risk for future SR. Recognizing the significance of frequent LLRs is important for designing safer protocols for successful SCIT.

In the Division of Allergy and Clinical Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, we performed SCIT in approximately 100 patients and 2000 injections per year. The LR associated SCIT were complained in 75% of the patients. Of the patients who experienced LR, 80% had LR more than 25 mm which was considered LLR.

Many strategies to prevent or minimize LR were reported. Oral antihistamines, leukotriene receptor antagonist (LTRA) or anti-IgE could reduce LR during the built-up phase. Cold compression or topical steroid were used to reduce the LR without any strong evidence. To our knowledge, the benefit of epinephrine coated syringe prior to drawing the allergen extract for SCIT in patients with frequent LLR has never been explored in any controlled trial.

The objective of this study is to compare the size of LR in patients with frequent LLR who receive SCIT by coating syringe with epinephrine or placebo prior to drawing allergen extract.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 6 years old who received SCIT at Pediatrics allergy departments at Siriraj hospital
* Patients who develops larges local reactions(mean wheal diameter > 25 mm.) during SCIT.
* Patients who received SCIT in maintenance phase.

Exclusion Criteria:

* Patients who develops systemic reactions (more than grade 1) during SCIT.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Epinephrine coated syringe for SCIT changed sized of large local reactions compared with placebo | 30 minutes, 2 hours, 4 hours, 6 hours
  We measured the sized of local reactions after injected SCIT coated with epinephrine or placebo for 30 minutes at clinic then 2 hours, 4 hours and 6 hours at home.

SECONDARY OUTCOMES:
Epinephrine coated syringe for SCIT changed systemic reactions compared with placebo. | 30 minutes, 2 hours, 4 hours, 6 hours
  We measured the systemic reactions after injected SCIT coated with epinephrine or placebo for 30 minutes at clinic then 2 hours, 4 hours and 6 hours at home.

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Orathai Piboonpocanun, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roy SR, Sigmon JR, Olivier J, Moffitt JE, Brown DA, Marshall GD. Increased frequency of large local reactions among systemic reactors during subcutaneous allergen immunotherapy. Ann Allergy Asthma Immunol. 2007 Jul;99(1):82-6. doi: 10.1016/S1081-1206(10)60626-6. PMID 17650835
- [Result] Calabria CW, Stolfi A, Tankersley MS. The REPEAT study: recognizing and evaluating periodic local reactions in allergen immunotherapy and associated systemic reactions. Ann Allergy Asthma Immunol. 2011 Jan;106(1):49-53. doi: 10.1016/j.anai.2010.10.025. PMID 21195945